CLINICAL TRIAL: NCT05751135
Title: Impact of Focal Muscle Vibration on Bio-psychosocial Outcomes in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-01289 KiranKhushnood
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Focal muscle vibration; Biopsychosocial; Functional near-infrared spectroscopy; Electroencephalography; Emotional reactivity
MeSH Terms: conditions — Cerebral Palsy | interventions — Resistance Training; Patient Positioning

STUDY DESIGN:
Intervention Model Description: 3 parallel group mixed methods
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focal muscle vibration group 1 (Experimental): Focal muscle vibration with frequency of 80 Hz will be provided 3 days along with stretching, strengthening and positioning for 8 weeks
  Interventions: Device: Focal muscle vibration; Procedure: Stretching; Procedure: Strengthening; Procedure: Positioning
- Focal muscle vibration group 2 (Experimental): Focal muscle vibration with frequency of 100 Hz will be provided 3 days a week along with stretching, strengthening and positioning for 8 weeks.
  Interventions: Device: Focal muscle vibration; Procedure: Stretching; Procedure: Strengthening; Procedure: Positioning
- Control group (Active Comparator): Stretching, strengthening and positioning in 3 sessions a week for 8 weeks
  Interventions: Procedure: Stretching; Procedure: Strengthening; Procedure: Positioning

INTERVENTIONS:
Device: Focal muscle vibration — Focal muscle vibration will be provided by a longitudinal muscle vibrator on muscles of lower limb; hamstrings, quadriceps, illiopsoas, calf, gluteus maximus and medius. Each muscle will be targeted 3 times with 30 seconds time period and keeping 10 second interval.
  Arms: Focal muscle vibration group 1; Focal muscle vibration group 2
Procedure: Stretching — Stretching of shortened lower extremity muscle
Procedure: Strengthening — Strengthening exercises for weak lower extremity muscles
Procedure: Positioning — Positioning of participant to maintain a good body posture

SUMMARY:
This study aims to determine the effects of focal muscle vibration on bio-psychosocial outcomes in subjects with cerebral palsy. Mixed methods will be used and the study will be conducted in 2 phases; 1st phase is determining the effects of intervention, whereas second step is prediction of outcomes. A qualitative gait analysis will also be done.

DETAILED DESCRIPTION:
The literature suggests the positive effects of focal muscle vibration on various motor components of cerebral palsy. Although there is a gap regarding it's effects with perspective of bio-psychosocial model, which will be the main focus of this study. The study will look for the effects of focal muscle vibration on biological, psychological and social aspects of subjects with cerebral palsy (CP). The intervention in form of focal muscle vibration and standard physical therapy will be provided for 12 weeks and the subjects will then be followed for 4 weeks to look for retention effects, and till 24 weeks for prediction of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed spastic diplegic cerebral palsy cases with following characteristics;
* Gross motor function classification scale levels II-IV
* Receiving standard physical therapy care

Exclusion Criteria:

* Severe cognitive, visual and hearing impairments.
* History of metabolic diseases.
* History of recent fractures.
* Children with severe musculo-skeletal anomalies

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy (fNIRS) | Baseline
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks.
Functional near-infrared spectroscopy (fNIRS) | After 4 weeks
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks.
Functional near-infrared spectroscopy (fNIRS) | After 8 weeks
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks.
Electroencephalogram (EEG) | Baseline
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention.
Electroencephalogram (EEG) | After 4 weeks
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention.
Electroencephalogram (EEG) | After 8 weeks
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention.
Gross Motor Function Measure | Baseline
  Gross motor function measure is a standard instrument which measures the change in motor function with time in CP subjects. It assess the amount of motor task a child can perform. an 88 point tool with scoring of 0-3 for each item, with 0 = doesn't initate activity to 3= complete the activity
Gross Motor Function Measure | After 4 weeks
  Gross motor function measure is a standard instrument which measures the change in motor function with time in CP subjects. It assess the amount of motor task a child can perform. an 88 point tool with scoring of 0-3 for each item, with 0 = doesn't initate activity to 3= complete the activity
Gross Motor Function Measure | After 8 weeks
  Gross motor function measure is a standard instrument which measures the change in motor function with time in CP subjects. It assess the amount of motor task a child can perform. an 88 point tool with scoring of 0-3 for each item, with 0 = doesn't initate activity to 3= complete the activity
Gross Motor Function Measure | After 12 weeks
  Gross motor function measure is a standard instrument which measures the change in motor function with time in CP subjects. It assess the amount of motor task a child can perform. an 88 point tool with scoring of 0-3 for each item, with 0 = doesn't initate activity to 3= complete the activity
Modified Ashworth scale | Baseline
  It is standard tool for measuring the spasticity with scoring 0-5, 0=no increase in muscle tone to 5=rigid in flexion and extension
Modified Ashworth scale | After 4 weeks
  It is standard tool for measuring the spasticity with scoring 0-5, 0=no increase in muscle tone to 5=rigid in flexion and extension
Modified Ashworth scale | After 8 weeks
  It is standard tool for measuring the spasticity with scoring 0-5, 0=no increase in muscle tone to 5=rigid in flexion and extension
Modified Ashworth scale | After 12 weeks
  It is standard tool for measuring the spasticity with scoring 0-5, 0=no increase in muscle tone to 5=rigid in flexion and extension
Child Behavior Checklist (CBCL) | Baseline
  The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioral problems in children and adolescents. There are 2 checklists; 1 for ages 1.5 to 5 years and other for 6 to 18 years of age.
Child Behavior Checklist (CBCL) | After 4 weeks
  The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioral problems in children and adolescents. There are 2 checklists; 1 for ages 1.5 to 5 years and other for 6 to 18 years of age.
Child Behavior Checklist (CBCL) | After 8 weeks
  The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioral problems in children and adolescents. There are 2 checklists; 1 for ages 1.5 to 5 years and other for 6 to 18 years of age.
Child Behavior Checklist (CBCL) | After 12 weeks
  The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioral problems in children and adolescents. There are 2 checklists; 1 for ages 1.5 to 5 years and other for 6 to 18 years of age.
Social support questionnaire | Baseline
  A 6 item questionnaire designed to measure perceptions of social support and satisfaction with that social support
Social support questionnaire | After 4 weeks
  A 6 item questionnaire designed to measure perceptions of social support and satisfaction with that social support
Social support questionnaire | After 8 weeks
  A 6 item questionnaire designed to measure perceptions of social support and satisfaction with that social support
Social support questionnaire | After 12 weeks
  A 6 item questionnaire designed to measure perceptions of social support and satisfaction with that social support
Self perception profile | Baseline
  Targeting the self-perception this tool is used to determine global psychosocial function and encompasses major domains; scholastic, social, athletic competence, physical appearance, behavioral conduct and global self-worth. There are 6 domains with 36 items in total with in each item is scored on a four-point scale from 1 to 4.
Self perception profile | After 4 weeks
  Targeting the self-perception this tool is used to determine global psychosocial function and encompasses major domains; scholastic, social, athletic competence, physical appearance, behavioral conduct and global self-worth. There are 6 domains with 36 items in total with in each item is scored on a four-point scale from 1 to 4.
Self perception profile | After 8 weeks
  Targeting the self-perception this tool is used to determine global psychosocial function and encompasses major domains; scholastic, social, athletic competence, physical appearance, behavioral conduct and global self-worth. There are 6 domains with 36 items in total with in each item is scored on a four-point scale from 1 to 4.
Self perception profile | After 12 weeks
  Targeting the self-perception this tool is used to determine global psychosocial function and encompasses major domains; scholastic, social, athletic competence, physical appearance, behavioral conduct and global self-worth. There are 6 domains with 36 items in total with in each item is scored on a four-point scale from 1 to 4.
Perth Emotional Reactivity Scale (PERS-S) | Baseline
  The Perth Emotional Reactivity Scale (PERS-S) is 18 item self-report measure of trait levels of emotional reactivity, derived from original version of 30 item.
Perth Emotional Reactivity Scale (PERS-S) | After 4 weeks
  The Perth Emotional Reactivity Scale (PERS-S) is 18 item self-report measure of trait levels of emotional reactivity, derived from original version of 30 item.
Perth Emotional Reactivity Scale (PERS-S) | After 8 weeks
  The Perth Emotional Reactivity Scale (PERS-S) is 18 item self-report measure of trait levels of emotional reactivity, derived from original version of 30 item.
Perth Emotional Reactivity Scale (PERS-S) | After 12 weeks
  The Perth Emotional Reactivity Scale (PERS-S) is 18 item self-report measure of trait levels of emotional reactivity, derived from original version of 30 item.
Modified Caregiver Strain Index (MCSI) | Baseline
  The Modified Caregiver Strain Index (MCSI) is used to screen for caregiver strain with long-term family caregivers. It is short and quick with 13 questions, which measures strain related to care provision.
Modified Caregiver Strain Index (MCSI) | After 4 weeks
  The Modified Caregiver Strain Index (MCSI) is used to screen for caregiver strain with long-term family caregivers. It is short and quick with 13 questions, which measures strain related to care provision.
Modified Caregiver Strain Index (MCSI) | After 8 weeks
  The Modified Caregiver Strain Index (MCSI) is used to screen for caregiver strain with long-term family caregivers. It is short and quick with 13 questions, which measures strain related to care provision.
Modified Caregiver Strain Index (MCSI) | After 12 weeks
  The Modified Caregiver Strain Index (MCSI) is used to screen for caregiver strain with long-term family caregivers. It is short and quick with 13 questions, which measures strain related to care provision.
Electromyography (EMG) | Baseline
  EMG will identify any changes in co-contraction between the muscles; quadriceps and hamstrings.
Electromyography (EMG) | After 4 weeks
  EMG will identify any changes in co-contraction between the muscles; quadriceps and hamstrings.
Electromyography (EMG) | After 8 weeks
  EMG will identify any changes in co-contraction between the muscles; quadriceps and hamstrings.
Trunk control measurement scale (TCMS) | Baseline
  Trunk control measurement scale will determine the level of trunk control in a child with CP. It comprises of static and dynamic sitting balance along with reaching activities which determine the equilibrium. The maximum score is 58, the higher the scores indicate better trunk control.
Trunk control measurement scale (TCMS) | After 4 weeks
  Trunk control measurement scale will determine the level of trunk control in a child with CP. It comprises of static and dynamic sitting balance along with reaching activities which determine the equilibrium. The maximum score is 58, the higher the scores indicate better trunk control.
Trunk control measurement scale (TCMS) | After 8 weeks
  Trunk control measurement scale will determine the level of trunk control in a child with CP. It comprises of static and dynamic sitting balance along with reaching activities which determine the equilibrium. The maximum score is 58, the higher the scores indicate better trunk control.
Trunk control measurement scale (TCMS) | After 12 weeks
  Trunk control measurement scale will determine the level of trunk control in a child with CP. It comprises of static and dynamic sitting balance along with reaching activities which determine the equilibrium. The maximum score is 58, the higher the scores indicate better trunk control.
Pediatric Balance Scale (PBS) | Baseline
  Pediatric Balance Scale will determine the level of balance and postural control in a child with CP. The maximum score is 56 and higher scores indicate better level of balance while score closer to zero indicate impaired balance.
Pediatric Balance Scale (PBS) | After 4 weeks
  Pediatric Balance Scale will determine the level of balance and postural control in a child with CP. The maximum score is 56 and higher scores indicate better level of balance while score closer to zero indicate impaired balance.
Pediatric Balance Scale (PBS) | After 8 weeks
  Pediatric Balance Scale will determine the level of balance and postural control in a child with CP. The maximum score is 56 and higher scores indicate better level of balance while score closer to zero indicate impaired balance.
Pediatric Balance Scale (PBS) | After 12 weeks
  Pediatric Balance Scale will determine the level of balance and postural control in a child with CP. The maximum score is 56 and higher scores indicate better level of balance, while score closer to zero indicate impaired balance.
Dynamometer | Bassline
  The dynamometer will be used to determine the strength in lower limb muscles; quadriceps, hamstrings, adductors and abductors of the CP subjects
Dynamometer | After 4 weeks
  The dynamometer will be used to determine the strength in lower limb muscles; quadriceps, hamstrings, adductors and abductors of the CP subjects
Dynamometer | After 8 weeks
  The dynamometer will be used to determine the strength in lower limb muscles; quadriceps, hamstrings, adductors and abductors of the CP subjects
Dynamometer | After 12 weeks
  The dynamometer will be used to determine the strength in lower limb muscles; quadriceps, hamstrings, adductors and abductors of the CP subjects
Cerebral Palsy Quality of Life (CPQOL) | Baseline
  Cerebral Palsy Quality of Life is tool to access the quality of life of children with CP it incorporates parental impact and family functioning along with concepts of illness, functional status, mental health, and comfort. Items are transformed to range of 0-100, the algebraic mean of item values is computer for each domain
Cerebral Palsy Quality of Life (CPQOL) | After 4 weeks
  Cerebral Palsy Quality of Life is tool to access the quality of life of children with CP it incorporates parental impact and family functioning along with concepts of illness, functional status, mental health, and comfort. Items are transformed to range of 0-100, the algebraic mean of item values is computer for each domain
Cerebral Palsy Quality of Life (CPQOL) | After 8 weeks
  Cerebral Palsy Quality of Life is tool to access the quality of life of children with CP it incorporates parental impact and family functioning along with concepts of illness, functional status, mental health, and comfort. Items are transformed to range of 0-100, the algebraic mean of item values is computer for each domain
Cerebral Palsy Quality of Life (CPQOL) | After 12 weeks
  Cerebral Palsy Quality of Life is tool to access the quality of life of children with CP it incorporates parental impact and family functioning along with concepts of illness, functional status, mental health, and comfort. Items are transformed to range of 0-100, the algebraic mean of item values is computer for each domain
Edinburgh Visual Gait Assessment Score | Baseline
  Edinburgh Visual Gait Assessment (EVGA) is an assessment tool which qualitatively asses various parameters of gait via video recordings. It uses lateral and anterior views of gait to identify the quality of gait patterns and movements.
Edinburgh Visual Gait Assessment Score | After 4 weeks
  Edinburgh Visual Gait Assessment (EVGA ) is an assessment tool which qualitatively asses various parameters of gait via video recordings. It uses lateral and anterior views of gait to identify the quality of gait patterns and movements.
Edinburgh Visual Gait Assessment Score | After 8 weeks
  Edinburgh Visual Gait Assessment Score (EVGA) is an assessment tool which qualitatively asses various parameters of gait via video recordings. It uses lateral and anterior views of gait to identify the quality of gait patterns and movements.
Edinburgh Visual Gait Assessment Score | After 12 weeks
  Edinburgh Visual Gait Assessment Score (EVGA) is an assessment tool which qualitatively asses various parameters of gait via video recordings. It uses lateral and anterior views of gait to identify the quality of gait patterns and movements.
Child friendly Depression Anxiety Stress Scale 21 (DASS-21) | Baseline
  A 21 item scale derive from DASS 42 to access the depression, anxiety and stress among children
Child friendly Depression Anxiety Stress Scale 21 (DASS-21) | After 4 weeks
  A 21 item scale derive from DASS 42 to access the depression, anxiety and stress among children
Child friendly Depression Anxiety Stress Scale 21 (DASS-21) | After 8 weeks
  A 21 item scale derive from DASS 42 to access the depression, anxiety and stress among children
Child friendly Depression Anxiety Stress Scale 21 (DASS-21) | After 12 weeks
  A 21 item scale derive from DASS 42 to access the depression, anxiety and stress among children
Immune Response Questionnaire (IRQ) | Baseline
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 6 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status
Immune Response Questionnaire (IRQ) | After 4 weeks
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 6 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status
Immune Response Questionnaire (IRQ) | After 8 weeks
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 6 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status
Immune Response Questionnaire (IRQ) | After 12 weeks
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and prolonged healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be repeated after 6 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status
Reaction Time | Baseline
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time
Reaction Time | After 4 weeks
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time
Reaction Time | After 8 weeks
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time
Reaction Time | After 12 weeks
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  It's a six-minute test that covers latency (response speed), correct responses and errors of commission and omission.
  More accurate reaction in less time inclines toward good reaction time
Heart rate variability (HRV) | Baseline
  Heart rate variability (HRV) will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual. Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders. Heart Rate will be monitored throughout the session. Assessment of participants will be continued throughout the intervention.
Heart rate variability (HRV) | After 4 weeks
  Heart rate variability (HRV) will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual. Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders. Heart Rate will be monitored throughout the session. Assessment of participants will be continued throughout the intervention
Heart rate variability (HRV) | After 8 weeks
  Heart rate variability (HRV) will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual. Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders. Heart Rate will be monitored throughout the session. Assessment of participants will be continued throughout the intervention
Heart rate variability (HRV) | After 12 weeks
  Heart rate variability (HRV) will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual. Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders. Heart Rate will be monitored throughout the session. Assessment of participants will be continued throughout the intervention
Manual Muscle Testing (MMT) | Baseline
  Manual muscle testing will be used to determine the strength of lower limb muscles. It has scores from 0 to 5, with 5 being the movement against maximum resistance and 0 being no contraction.
Manual Muscle Testing (MMT) | After 4 weeks
  Manual muscle testing will be used to determine the strength of lower limb muscles. It has scores from 0 to 5, with 5 being the movement against maximum resistance and 0 being no contraction.
Manual Muscle Testing (MMT) | After 8 weeks
  Manual muscle testing will be used to determine the strength of lower limb muscles. It has scores from 0 to 5, with 5 being the movement against maximum resistance and 0 being no contraction.
Manual Muscle Testing (MMT) | After 12 weeks
  Manual muscle testing will be used to determine the strength of lower limb muscles. It has scores from 0 to 5, with 5 being the movement against maximum resistance and 0 being no contraction.
Semi structured interview | After 8 weeks
  A semi-structured interview will be conducted with parents/ caregivers of CP subjects focusing on the feedback about treatment protocols and social, psychological and physical status and needs, and any observed change in needs or status

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University; Kiran Khushnood, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Al-Farabi Special Education Center For (P.H.C), Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No